CLINICAL TRIAL: NCT07144813
Title: Clinical Post- Approval Study of the Neuspera Sacral Neuromodulation (SNM) System in Patients With Symptoms of Urinary Urgency Incontinence (UUI)
Brief Title: Post-Approval Study of the Neuspera Sacral Neuromodulation System
Acronym: NSM-005
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuspera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neuspera Medical (NSM-005)
Record Dates: First submitted 2025-08-25; First posted 2025-08-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Urinary Urgency Incontinence
Keywords: UUI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Neuspera Implantable Sacral Neuromodulation Stimulation System (Other): Long term follow-up for the FDA approved Neuspera Sacral Neuromodulation Stimulation system
  Interventions: Device: Neuspera Implantable Sacral Neuromodulation System

INTERVENTIONS:
Device: Neuspera Implantable Sacral Neuromodulation System — Stimulation of the Sacral Nerve.

SUMMARY:
Prospective, multi-center, single-arm, post-approval study is designed to assess the long-term safety and efficacy data of the Neuspera Sacral Neuromodulation (SNM) System following commercial approval of the Neuspera SNM System.

Participants in this study received intervention/implanted in Phase I or Phase II of the Neuspera SANS_UUI (NSM-004) Study.

DETAILED DESCRIPTION:
The Neuspera SNM System received FDA PMA approval for the treatment of urinary urge incontinence in subjects who have failed, could not tolerate, or were not a candidate for more conservative treatment. The study will serve as the Post Approval Study (PAS) requirement of the PMA Approval.

This post approval study (PAS) is designed to assess the long-term safety and effectiveness data out to 72 months post-implant, in consenting subjects implanted in Phase I or Phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the SANS-UUI Phase I or Phase II study

Exclusion Criteria:

* None

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Through 72 months
  Incidence of device- and procedure-related AEs
Primary Effectiveness Endpoint: | Through 72 months
  Percentage of all implanted subjects who experience an improvement in UUI episodes of at least 50% or more

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Padron, MD, Principal Investigator — Florida Urology Partners
Locations (20):
- United States (20):
  - Kaiser Permanente Point Loma MOB, San Diego, California
  - Genesis Healthcare Partners, San Diego, California
  - Florida Urology Partners, Tampa, Florida
  - Women's Health Advantage,, Fort Wayne, Indiana
  - Indiana University, School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center,, Kansas City, Kansas
  - University of Louisville Health System,, Louisville, Kentucky
  - Ochsner Medical, New Orleans, Louisiana
  - University of Michigan Health, Wyoming, Michigan
  - Minnesota Urology, Woodbury, Minnesota
  - Specialty Research of St. Louis, St Louis, Missouri
  - Adult & Pediatric Urology P.C, Omaha, Nebraska
  - Premier Medical Group,, Poughkeepsie, New York
  - MetroHealth System,, Cleveland, Ohio
  - Women's Healthcare Associates,, Portland, Oregon
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery,, North Wales, Pennsylvania
  - Southern Urogynecology,, West Columbia, South Carolina
  - Urology Austin,, Austin, Texas
  - UCNT Dallas,, Dallas, Texas
  - Virginia Mason Medical Center,, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuspera Medical web page — http://neuspera.com